CLINICAL TRIAL: NCT00634855
Title: Endothelial Progenitor Cells in Umbilical Cord Blood in Preeclampsia and IUGR
Status: Terminated | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Ashley Ryan, MD, Medical University of South Carolina
Other Study IDs: HR # 17821
Record Dates: First submitted 2008-02-19; First posted 2008-03-13 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Preeclampsia; IUGR
Keywords: Endothelial progenitor cells; Endothelial dysfunction
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Complicated: Women with pregnancies complicated by intrauterine growth restriction or preeclampsia
- Normal: Women with normal pregnancies

SUMMARY:
The objective of this study is to determine whether there are alterations in the population of endothelial progenitor cells in umbilical cord blood samples of infants born in the setting of maternal preeclampsia or fetal growth restriction.

DETAILED DESCRIPTION:
Preeclampsia remains a significant cause of neonatal and maternal morbidity and mortality. This disorder is found in 5-7% of pregnancies and its incidence is increased in gravid patients with multiple gestations, chronic hypertension, renal disease, autoimmune disease, and at extremes of maternal age. It is responsible for 15% of preterm births which is accompanied by a resultant increase in neonatal morbidity and mortality. In developing countries, it is responsible for approximately 50,000 maternal deaths each year. No widespread intervention to prevent this disease has been found effective and the only effective treatment remains delivery of the fetus.

To date, the cause of preeclampsia is not known although many agree that preeclampsia is a two-stage disease as described by Roberts et al. with the placenta of central importance. The first stage involves poor placental perfusion usually a result of impaired vascular remodeling in early pregnancy or from maternal disease. This leads to the second stage, which is the maternal syndrome of preeclampsia and involves both endothelial and leukocyte activation.

Preeclampsia is associated with an increased maternal cardiovascular risk later in life. Women with a history of preeclampsia demonstrate altered expression of angiogenesis-related proteins and increased insulin resistance as measured by the homeostasis model of insulin resistance. Additionally, preeclampsia is associated with an increase in future cardiovascular risk in the fetus.

Endothelial dysfunction and abnormal regulation of vascular tone that is present in preeclampsia suggests abnormal development of vascular cells such as endothelial progenitor cells. The increased cardiovascular risk of neonates born in the setting of IUGR and preeclampsia also suggests the possibility of abnormal development of endothelial progenitor cells in the fetal compartment in these disease states. The purpose of this pilot project is to determine the effects of preeclampsia/IUGR on endothelial progenitor cells derived from fresh umbilical cord blood.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18-45
* Gestational age between 30-40 weeks plus:

  * Uncomplicated pregnancy or
  * Fetal estimated weight <10% for gestational age or abdominal circumference <5% or
  * Preeclampsia by ACOG criteria:

    1. HTN > 140/90 on two occasions
    2. Proteinuria > 300mg on 24 hour urine specimen or 1+ on urine dip

Exclusion Criteria:

* Non-reassuring fetal status
* Congenital abnormalities
* Multiple gestations
* Clinical Chorioamnionitis
* Recent infectious disease (within 2 weeks)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women who are between 30 and 40 weeks gestation and are admitted to MUSC.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Proportions of endothelial progenitor cells present in umbilical cord | After birth

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Ryan, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States